CLINICAL TRIAL: NCT07260201
Title: Evaluating the Triglyceride-Glucose Index and TGI-BMI for Insulin Resistance Assessment: A Comparative Study With HOMA-IR
Brief Title: Triglyceride-Glucose and TGI-BMI Indices Compared With HOMA-IR
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Bekir Sami Uyanık, Professor of Clinical Biochemistry, Hisar Intercontinental Hospital, Hisar Intercontinental Hospital
Other Study IDs: HIH 2025 HOMA IR
Record Dates: First submitted 2025-11-18; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Insulin Resistance; Obesity Type 2 Diabetes Mellitus
Keywords: Insulin resistance; Triglyceride-glucose index; TGI-BMI; HOMA-IR
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group/Cohort 1 Label: Non-Insulin Resistant (Non-IR) Group: Group 1 - Non-Insulin Resistant (Non-IR) Group
  Participants with HOMA-IR values below 2.5, classified as non-insulin resistant. Anthropometric and biochemical data (including fasting glucose, triglycerides, and BMI) were analyzed retrospectively to calculate TGI and TGI-BMI indices.
- Group/Cohort 2 Label: Insulin Resistant (IR) Group: Group 2 - Insulin Resistant (IR) Group
  Participants with HOMA-IR values greater than 2.5, classified as insulin resistant. Anthropometric and biochemical measurements were reviewed from medical records, and TGI and TGI-BMI indices were compared with those of the Non-IR group.

SUMMARY:
Insulin resistance plays a key role in the development of type 2 diabetes, metabolic syndrome, and heart disease. The most common way to measure insulin resistance is the HOMA-IR index, but it requires fasting insulin tests, which are not always available in clinical practice.

This study aims to assess two simpler and more accessible alternatives: the triglyceride-glucose index (TGI) and its body mass index-adjusted version (TGI-BMI). Data from 150 adult patients were analyzed retrospectively and divided into groups according to their insulin resistance status. Standard laboratory and body measurements were compared between groups, and statistical analyses were used to determine how well TGI and TGI-BMI identify insulin resistance.

The results showed that both TGI and TGI-BMI were closely related to insulin resistance and demonstrated high diagnostic accuracy, similar to HOMA-IR. The TGI-BMI index was particularly effective in individuals with obesity. These findings suggest that TGI and TGI-BMI could serve as practical, low-cost alternatives to HOMA-IR for evaluating insulin resistance in clinical and population settings where insulin testing is not routinely available.

DETAILED DESCRIPTION:
Insulin resistance (IR) is a central feature of metabolic and cardiovascular disorders, yet the routine measurement of fasting insulin required for HOMA-IR limits its clinical applicability. The triglyceride-glucose index (TGI) and its body mass index-adjusted form (TGI-BMI) have emerged as simple, cost-effective surrogates that rely only on standard biochemical data.

This retrospective study analyzed data from 150 adults evaluated at Hisar Intercontinental Hospital. Participants were categorized into insulin-resistant (HOMA-IR > 2.5) and non-resistant (HOMA-IR < 2.5) groups. Anthropometric and biochemical variables were obtained from medical records. TGI and TGI-BMI values were calculated for each participant, and comparisons were made between groups. Correlation and receiver operating characteristic (ROC) analyses were used to determine the relationship and diagnostic accuracy of these indices relative to HOMA-IR.

The study aims to validate TGI and TGI-BMI as reliable, low-cost indicators of insulin resistance applicable in both clinical and epidemiological settings, especially in laboratories where insulin assays are unavailable. The findings may contribute to improved screening and risk assessment strategies in metabolic disease management.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were adults aged 18-65 years with complete fasting biochemical and anthropometric data. Only patients who were not receiving antidiabetic medications at the time of evaluation were included.

Exclusion Criteria:

* Patients were excluded if they had any of the following:

  * Known endocrine disorders (e.g., thyroid dysfunction, Cushing's syndrome)
  * Chronic kidney or liver disease
  * Active infection or systemic inflammatory disease
  * Ongoing use of medications known to affect glucose or lipid metabolism (e.g., corticosteroids, statins, metformin, or insulin)
  * Incomplete or missing laboratory data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent routine biochemical testing and metabolic evaluation at Hisar Intercontinental Hospital. Data were obtained retrospectively from medical records. Participants were divided into two cohorts based on insulin resistance status determined by HOMA-IR values:
  Non-Insulin Resistant (HOMA-IR < 2.5)
  Insulin Resistant (HOMA-IR > 2.5)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the Triglyceride-Glucose Index (TGI) for detecting insulin resistance | Retrospective data analysis (single time point).
  Area under the receiver operating characteristic (ROC) curve (AUC), sensitivity, and specificity of TGI in identifying insulin resistance compared to HOMA-IR (>2.5 as reference).

SECONDARY OUTCOMES:
Diagnostic accuracy of the BMI-adjusted Triglyceride-Glucose Index (TGI-BMI) | Retrospective data analysis (single time point).
  ROC curve analysis of TGI-BMI compared with HOMA-IR; AUC, sensitivity, specificity values recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Bekir Sami Uyanık, MD, Prof, Principal Investigator — Hisar Intercontinental Hospital; Selami Aydin, MD, Study Director — Hisar Intercontinental Hospital; Süleyman İpekci, Prof, Study Chair — Hisar Intercontinental Hospital and Atlas University
Locations (1):
- Hisar Intercontinental Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Participant data (PD) and supporting information will be available starting from the date of publication of the study results. The data will remain accessible for a period of 5 years after publication.
Access Criteria: Access to the Individual Participant Data (IPD) and supporting information will be limited to authorized members of the study team and independent researchers who submit a formal request for scientific evaluation. Accessible materials will include the de-identified IPD dataset, study protocol, and relevant analysis outputs
URL: https://hisarhospital.com/doktorlarimiz/prof-dr-bekir-sami-uyanik/

REFERENCES:
- See also: This publication supports the present study by demonstrating that the triglyceride-glucose (TyG) index is independently associated with an increased risk of diabetes, even among individuals with normal fasting triglyceride and glucose levels. It provides — https://pubmed.ncbi.nlm.nih.gov/40589514/
- Available data/document: Individual participant data will not be shared because the study is retrospective and based on anonymized medical records.: no identifier available — https://www.hisarhospital.com — This publication provides background evidence supporting the evaluation of triglyceride-glucose-based indices as markers of insulin resistance.